CLINICAL TRIAL: NCT01867840
Title: Study of the Role of Acid Sensing Ion Channels (ASICs) in Human Inflammatory Pain
Brief Title: Role of ASICs in Human Inflammatory Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 12-PP-07
Record Dates: First submitted 2013-05-15; First posted 2013-06-04 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Arthritis; Osteoarthritis; Chondrocalcinosis; Gouty Arthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis; Osteoarthritis; Chondrocalcinosis; Arthritis, Gouty; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (1):
- arthritis

SUMMARY:
In recent years, ion channels have emerged as new therapeutic targets for pain. Among these channels, ASICs (Acid Sensing Ion Channels) are of particular interest because they are directly activated by extracellular acidity, which is a major cause of pain. Indeed, many painful conditions such as ischemia, inflammation, tumor development or tissue incision are accompanied by tissue acidification. ASIC are excitatory ion channels that are expressed in neurons, including nociceptive sensory neurons. In humans, the use of amiloride, a nonspecific inhibitor of ASICs, has demonstrated their role in the perception of pain induced by subcutaneous injections of acidic solutions. ASICs thus appear as new candidates capable of mediating pain in humans. A growing number of data suggests that, in addition to protons, ASICs may also be activated by one or more endogenous compounds produced during inflammation. The purpose of this research project is to identify these compounds by testing the effects of human inflammatory exudates on ASICs activity. The discovery of such compounds would definitely validate ASICs as novel therapeutic targets for pain treatment in humans

ELIGIBILITY:
Inclusion Criteria:

* septic arthritis
* gonarthrosis in push-inflammatory
* microcrystalline arthropathies
* chronic inflammatory rheumatism

Exclusion Criteria:

* refusal to participate in the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: (osteoarthritis, chondrocalcinosis, gouty arthritis, rheumatoid arthritis)
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
activation or miodulation to Electrical potential of ionic channel in the synovial fluid | 1 day
  only once because it's an single ponction of sinovial fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique BREUIL, Pr, Principal Investigator — service de rhumatologie
Locations (1):
- Service de Rhumatologie, Nice, Nice, France

REFERENCES:
- [Derived] Khoury S, Colas J, Breuil V, Kosek E, Ahmed AS, Svensson CI, Marchand F, Deval E, Ferreira T. Identification of Lipid Biomarkers for Chronic Joint Pain Associated with Different Joint Diseases. Biomolecules. 2023 Feb 9;13(2):342. doi: 10.3390/biom13020342. PMID 36830710